CLINICAL TRIAL: NCT00617071
Title: Tailored Navigation in CRC Screening
Brief Title: Personalized Screening Plans to Increase Colorectal Cancer Screening in Healthy Participants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Health Services Research
Other Study IDs: CDR0000584278; TJUH-2006-44
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Occult Blood

INTERVENTIONS:
Other: medical chart review
Other: survey administration
Procedure: fecal occult blood test
Procedure: screening colonoscopy

SUMMARY:
RATIONALE: Developing a personalized screening plan may be more effective than usual care in increasing the number of healthy participants who regularly undergo screening for colorectal cancer.

PURPOSE: This randomized phase III trial is studying personalized screening plans to see how well they work compared with usual care in increasing colorectal cancer screening in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the impact of tailored intervention vs standard intervention vs usual care on patient utilization of colorectal cancer (CRC) screening.
* To compare the impact of these interventions on CRC screening preference.
* To compare the impact of these interventions on patient perceptions about CRC screening.

OUTLINE: This is a multicenter study. Participants are stratified by practice and study wave and blocking. Participants are randomized to 1 of 3 arms.

* Arm I (usual care): Participants receive usual care in accordance with their normal patterns of interaction with study practices.
* Arm II (standard intervention [SI]): A generic screening invitation letter, a colorectal cancer (CRC) screening informational booklet, stool blood testing (SBT) cards, and instructions for arranging a colonoscopy screening appointment are mailed to participants on day 15. On day 45, a reminder letter is mailed to participants who have not completed SBT or undergone a screening colonoscopy.
* Arm III (tailored navigation intervention [TNI]): A test-specific screening invitation letter, a CRC screening informational booklet, and additional test-specific materials (i.e., instructions for arranging a colonoscopy screening appointment or SBT cards) are mailed to participants on day 15. On day 30, a patient navigator contacts participants by telephone who have not completed SBT or undergone a screening colonoscopy. The patient navigator re-assesses screening test-specific decision stage; addresses CRC screening barriers; develops a personalized CRC screening plan to move the participant towards screening use (i.e., explains the steps in completing the SBT or scheduling a colonoscopy appointment); and facilitates screening plan implementation. On day 45, a reminder letter is mailed to participants who were contacted by the navigator.

Participants in all arms complete a survey at baseline and then at 6 months. Medical records for each participant are reviewed at 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets the following criteria:

  * No personal history of colorectal neoplasia (cancer or polyps) or inflammatory bowel disease
  * No family history of colorectal cancer (CRC) diagnosed before the age of 60
  * Visited one of the six community-based primary care practices that are part of the Christiana Care Health System (CCHS) in Delaware within the past 2 years
  * Not up-to-date with CRC screening, according to the United States Preventive Services Task Force guidelines

PATIENT CHARACTERISTICS:

* Must have a complete address and telephone number
* Able to communicate in English
* No psychosis or severe dementia

PRIOR CONCURRENT THERAPY:

* No prior participation in the developmental study CA10241

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Screening utilization over the 6-month observation period

SECONDARY OUTCOMES:
Screening preference
Perceived salience and coherence and self-efficacy related to colorectal cancer (CRC) screening
Number and length of contacts with each participant and the type of communication during those contacts
Identification of predictors of CRC screening use and screening preference

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Myers, PhD, Study Chair — Jefferson Medical College of Thomas Jefferson University
Locations (1):
- Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania, United States